CLINICAL TRIAL: NCT00629577
Title: Ex Vivo Gene Expression Profiling of Cervical Cancer Progression in Biopsies And Tissue Samples From Patients With Cervical Lesions
Brief Title: Gene Expression Profiling of Cervical Cancer Progression in Biopsies and Tissue Samples
Acronym: SAGE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: no funding
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000581308; R01CA103830 (NIH); BCCR-H05-60100 (Other: UBC-BCCA REB)
Record Dates: First submitted 2008-03-05; First posted 2008-03-06 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2010-11

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Microarray Analysis; Flow Cytometry; Biopsy; Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: microarray analysis
Other: flow cytometry
Procedure: biopsy
Procedure: colposcopy

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial is studying gene expression profiling of cervical cancer progression in biopsies and tissue samples from patients with cervical lesions.

DETAILED DESCRIPTION:
OBJECTIVES:

* Classify cervical cancer progression at a molecular level using gene expression profiling generated from expression microarrays.
* Profile gene expression changes of dysplasia and early carcinoma of uterine cervical tissue at a molecular level using expression microarrays.
* Define a set of genes that classify the various grades of cervical cancer/dysplasia at a molecular level.
* Compare the expression profiles of clinical data to determine how accurately cell lines model the in vivo environment.

OUTLINE: Patients undergo colposcopy and a cervical smear is taken for flow cytometry analysis. Patients also undergo 2 biopsies from one clinically abnormal or normal site. Tissue samples are analyzed by gene expression profiling using human expression microarrays containing approximately 40,000 unique sequences. Data analysis consists of defining a set of genes, containing new targets for biomarkers, that classify the biopsies into 3 grades.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically suspicious malignant or premalignant cervical lesion

Criteria

Inclusion criteria:

* Included subjects will be ≥18 years old.
* Included subjects will not be pregnant.
* Included subjects will have a negative urine pregnancy test.
* Included subjects will be scheduled for colposcopy and/or LEEP treatment at the VGH Women's Clinic.
* Included subjects will indicate understanding of the study.
* Included subjects will provide informed consent to participate.

Exclusion criteria:

* Individuals <18 years old will be excluded.
* Pregnant individuals will be excluded.
* Individuals that have had an operation to remove their cervix will be excluded.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Classification of cervical cancer progression at a molecular level using gene expression profiling
Gene expression changes by microarray
Set of genes that classify the various grades of cervical cancer/dysplasia
Comparison of the expression profiles of clinical data to determine how accurately cell lines model the in vivo environment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Ehlen, M.D., Principal Investigator — BC Cancer Agency, Vancouver General Hospital
Locations (1):
- BC Cancer Research Centre, Vancouver, British Columbia, Canada